CLINICAL TRIAL: NCT03463434
Title: A Randomized Controlled Pilot Study Comparing Air Fluidized Therapy (AFT) to a Continuous Low Pressure (CLP) Low Air Loss (LAL) Support Surface in the Treatment of Stage 3 or 4 Pressure Injuries
Brief Title: AFT/CLP-LAL RCT Stage 3 or 4 Pressure Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hill-Rom (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR-SS2017-007
Record Dates: First submitted 2018-02-26; First posted 2018-03-13 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2018-09

CONDITIONS: Pressure Ulcer
Keywords: pressure ulcer treatment; wound healing
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: This multi-center, randomized, open-label, two treatment, parallel group study is designed to obtain comparative data on the healing rates of type 3 & 4 pressure injuries.
  The randomization schedule will be set up in blocks, and within a block, the randomization numbers will be assigned equally to the two treatment groups (Envella AFT, FIS bed surface types). A separate randomization schedule will be set up for each stage (3, 4 PI). The anticipated number of investigative sites is 3.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Air Fluidized Therapy (Experimental): Patients will be placed on the Envella AFT bed
  Interventions: Device: Air Fluidized Therapy
- Continuous Low Pressure-LAL (Active Comparator): Patients will receive a Continuous low pressure mattress with low air loss
  Interventions: Device: Continuous Low Pressure-LAL

INTERVENTIONS:
Device: Air Fluidized Therapy — AFT bed used for pressure injury treatment
  Arms: Air Fluidized Therapy
Device: Continuous Low Pressure-LAL — Continuous Low Pressure/Low Air Loss Mattress for Pressure injury treatment
  Arms: Continuous Low Pressure-LAL

SUMMARY:
Patients who have at least one stage 3 or 4 PI and are admitted to a participating treating facility will be candidates for study enrollment. Patients must provide written informed consent. Standard care for their admitted condition will be provided for the patients except for support surface selection, laboratory blood tests, PI measurement(s) by the 3-D camera measurement tool, and added pain and patient satisfaction assessments. Clinical assessments will be recorded weekly as described below. Patients will be followed until discharge from the LTACH or until 1) they require a different mattress for their admitted condition; or 2) reach a maximum of 12 weeks in the LTACH. At study discontinuation, a clinical general assessment of the quality of improvement of the PIs will be recorded.

DETAILED DESCRIPTION:
Patients admitted to the LTACH with at least one stage 3 or 4 PI will be evaluated for possible inclusion/exclusion criteria. Patients will be approached by the investigator, or their designee to acquire patient informed consent. If provided, patients will be randomized to their designated support surface, the bed will be ordered and patients will begin the study with a baseline study visit (week 0) that will include:

* Date and time of study bed placement
* A brief medical history, that includes current diagnoses, assessment of co-morbidities, an assessment of neurologic status, nutritional status, level of mobility, history of current PI's, documentation of treatments that have been applied to PI(s) prior to study entry
* Braden PU risk assessment (overall and subscores)
* Assessment of pain associated with the PI using a pain numeric rating scale (NRS), where patients rate their current pain intensity from 0 ("no pain") to 10 ("worst possible pain") [21]
* Blood for CBC, Albumin, Pre-Albumin, CRP will be collected.
* PI assessments: all PI's located on the lower truncal region of the patient's body will be assessed both subjectively by the treating clinicians for clinical signs of infection, as well as by a 3D wound assessment tool.
* Overall health status assessment

Subsequent weekly study visits will continue for a maximum of 12 weeks. The interim study visit documentation will include:

* Overall health status assessment of health (whether the patient's health is improving, maintaining, or worsening)
* Skin assessment to document any new PI's that may have developed,
* Braden PU risk assessment (overall and subscores)
* 3D Wound assessments of all lower truncal PI's,
* Clinical Assessment of signs and symptoms of wound infection
* Confirmation of support surface type,
* Documentation of adverse device effects, device-related complaints (within 24 hours of effect/complaint).

Clinical Resource Utilization Data: documentation of the following data will aim to achieve estimated clinical resources associated with caring for PIs:

* Documentation of dressing supplies,
* Debridement method, duration and frequency
* Type of antibiotics dosage, frequency, and duration
* Other pharmacologic agents used for wounds with dosage, frequency, and duration
* Assessment of pain
* Rental bed cost estimates
* Documentation of professional healthcare visits and/or types of healthcare services in the preceding week.
* Documentation of acute care hospitalizations
* An estimate of LTACH staff time devoted to wound care per day for that study week.

At study discharge, which may occur at the time of study PI healing, LTACH discharge, or upon stepdown from the randomized study surface) or for other reasons, a final study visit will be completed that includes:

* Date and time of study bed removal
* Overall health status assessment,
* Skin assessment to document any new PI's that may have developed,
* Braden PU risk assessment (includes subscores),
* 3D wound assessments of all truncal PI's,
* Clinical assessment of signs and symptoms of wound infection
* Confirmation of bed support surface type
* Documentation of adverse device effects, device related complaints (within 24 hours of effect/complaint).
* Clinical Resource Utilization Data:

  * documentation of dressing supplies,
  * debridement method, duration and frequency
  * type of antibiotics, dosage, frequency, and duration
  * other pharmacologic agents used for wounds with dosage, frequency, and duration,
  * rental bed cost estimates
  * documentation of professional healthcare visits and/or types of healthcare services in the preceding week.
  * documentation of acute care hospitalizations
  * an estimate of LTACH staff time devoted to wound care per day for that study week.
* Assessment of pain
* A patient bed satisfaction assessment will be completed if the patient is able to communicate
* Blood for CBC, Albumin, Pre-Albumin, CRP will be collected

ELIGIBILITY:
Inclusion Criteria:

1. Patient's treatment goals are curative or maintaining, and not palliative in nature.
2. Patient is compliant with standard clinical care for their admitted condition.
3. Patient's age is between 18 and 85 years
4. Patient is expected to have at least a 3-4-week length of stay (from date of assessment) in the treating LTACH
5. Patient must have at least one stage 3 or 4 PI located on the weight bearing aspect of the patient's truncal /pelvic region
6. Patients or their legal authorized representative must be willing and able to provide written informed consent.

Exclusion Criteria:

1. Patient has an unstable spinal cord injury
2. Patient weighs less than 70 lbs or more than 350 lbs.
3. The primary study PI site has had previous flaps or grafts with significant associated scarring which is clinically thought to impede wound contracture.
4. Patients with PIs where bone exposure is > 2 cm2 in area.
5. Patients with active osteomyelitis (via clinical assessment) or patients who have been diagnosed with osteomyelitis and have not yet completed a 6-8-week course of antibiotics
6. The primary study PI is located over the trochanteric head of the femur.
7. Patients that are currently taking or have taken in the last 6 weeks chemotherapy which is known to be cyto-toxic, or anti-angiogenic
8. Patients currently require immune modulating drugs (Humira (alalimumab), Orencia (abatacept), etc.)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2019-08-14 (Actual); Study Completion 2019-08-14 (Actual)

PRIMARY OUTCOMES:
Pressure ulcer healing | up to 12 weeks
  Volume (mm3)

SECONDARY OUTCOMES:
New Pressure Ulcers | up to 12 weeks
  new pressure ulcers
Length of stay | up to a year
  Length of stay in the Long-term Acute Care Hospital

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Noland Health Anniston, Anniston, Alabama
  - Noland Health, Birmingham, Alabama

IPD SHARING:
Plan to Share IPD: Undecided